CLINICAL TRIAL: NCT02892513
Title: Auricular Percutaneous Electrical Nerve Field Stimulation for Postoperative Pain Control in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Carrie Peterson, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00027872
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative
Keywords: Colorectal Surgery; transcutaneous electric nerve stimulation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Stimulation (Experimental): Participants will have active percutaneous auricular neurostimulation for 5 days during and after elective surgery.
  Interventions: Device: Percutaneous auricular neurostimulation
- Sham Percutaneous Neurostimulation (Sham Comparator): Participants will have inactive device worn for 5 days during and after elective surgery.
  Interventions: Device: Sham percutaneous auricular neurostimulation

INTERVENTIONS:
Device: Percutaneous auricular neurostimulation — The Bridge device (manufactured by Key Electronics [Jeffersonville, IN, USA] and distributed by Innovative Health Solutions [Versailles, IN, USA]) provides continual neurostimulation for five days with alternating current.
  Arms: Active Stimulation
Device: Sham percutaneous auricular neurostimulation — Identical in appearance to active, device, but no stimulation will be given.
  Arms: Sham Percutaneous Neurostimulation

SUMMARY:
Pain after surgery is unavoidable, and opioid medications are the cornerstone of most pain management regimens. However, they come at a cost with profound impacts on gastrointestinal motility, respiratory depression, and even long-term dependence. Stimulating the external ear with cutaneous electrical current is similar to acupuncture and could help improve postoperative pain. The Bridge device (manufactured by Key Electronics [Jeffersonville, IN, USA] and distributed by Innovative Health Solutions [Versailles, IN, USA]), has been used with success in treating opioid withdrawal and in animal studies has shown increases in pain thresholds. The investigators propose a prospective, randomized, placebo-controlled, double-blinded trial to evaluate if auricular neurostimulation improves postoperative pain and reduces opioid requirements for patients undergoing elective colon surgery.

pain perception in post-operative patients may be modulated via the auricular branch of the vagus nerve. This has the potential to reduce the use of opioid medications, which will in turn reduce the incidence of postoperative ileus and reduce patient need for and dependence on narcotic pain medications. This would have an enormous economic impact due to decreased length of hospital stays for patients who undergo abdominal surgery. In addition, opioid reduction could potentially lessen the national crisis of opioid addiction.

ELIGIBILITY:
Inclusion Criteria:

* elective colon surgery
* age over 18 years
* provide informed consent

Exclusion Criteria:

* emergency surgery
* history of opioid dependence/use, anxiety with anxiolytic use
* planned ICU admission postoperatively
* adhesive allergy/sensitivity
* other medical contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-11; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Blank JJ, Liu Y, Yin Z, Spofford CM, Ridolfi TJ, Ludwig KA, Otterson MF, Peterson CY. Impact of Auricular Neurostimulation in Patients Undergoing Colorectal Surgery with an Enhanced Recovery Protocol: A Pilot Randomized, Controlled Trial. Dis Colon Rectum. 2021 Feb 1;64(2):225-233. doi: 10.1097/DCR.0000000000001752. PMID 33417346

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Participants will have active percutaneous auricular neurostimulation for 5 days during and after elective surgery.
  Percutaneous auricular neurostimulation: The Bridge device (manufactured by Key Electronics [Jeffersonville, IN, USA] and distributed by Innovative Health Solutions [Versailles, IN, USA]) provides continual neurostimulation for five days with alternating current.
- Inactive: Participants will have inactive device worn for 5 days during and after elective surgery.
  Sham percutaneous auricular neurostimulation: Identical in appearance to active, device, but no stimulation will be given.
Period: Overall Study
Arm/Group | Active | Inactive
Started | 28 | 25 (did not receive allocated intervention = 1 (withdrew per participant request))
Completed | 28 (Discontinued intervention early = 5; excluded from analysis = 0) | 24 (Discontinued intervention early = 6; excluded from analysis = 1)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Inactive | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant withdrew before device was applied and data not collected for analysis
  years
    number analyzed (Participants) | 28 | 24 | 52
    (all) | 56.05 (11.266) | 61.49 (11.273) | 58.77 (11.248)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant withdrew before device was applied and data not collected for analysis
  Participants
    number analyzed (Participants) | 28 | 24 | 52
    Female | 14 | 9 | 23
    Male | 14 | 15 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: 1 participant withdrew before device was applied and data not collected for analysis
  participants
    United States: number analyzed (Participants) | 28 | 24 | 52
    United States | 28 | 24 | 52
Open vs Laparoscopic Technique [Count of Participants; unit: Participants] — Population: 1 participant withdrew before device was applied and data not collected for analysis
  Participants
    number analyzed (Participants) | 28 | 24 | 52
    Open | 2 | 7 | 9
    Laparoscopic | 26 | 17 | 43

OUTCOME MEASURES:

1. Primary Outcome: Total Narcotic Consumption During Hospital Stay
Description: Total inpatient narcotic use measured in oral morphine equivalents per day (OME)
Time Frame: 5 days
Population: 1 participant withdrew before device was applied and data not collected for analysis.
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalents per day (OME)
Arm/Group | Active | Inactive
Number analyzed (Participants) | 28 | 24
Oral Morphine Equivalents per day (OME) | 90.79 (54.93) | 90.30 (43.03)
Statistical Analysis 1: Comparison: Active vs Inactive; Test type: Superiority; p = 0.97, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Active | Inactive
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/24
Other Adverse Events (participants affected / at risk) | 0/28 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=28) | Inactive (N=24)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
GI Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02892513/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02892513/SAP_001.pdf
  • Informed Consent Form (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT02892513/ICF_002.pdf